CLINICAL TRIAL: NCT06901024
Title: Investigation of the Effects of Neuromobilization, Tendon Gliding, and Robotic Glove-Assisted Exercises on Pain, Grip Strength, and Hand Function in Patients With Hand Osteoarthritis
Brief Title: Effects of Neuromobilization, Tendon Gliding, and Robotic Glove-Assisted Exercises on Hand Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Head of Physiotherapy Department, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/081
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Neuromobilization; Tendon gliding; Robotic Assistive Device
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: The patients were divided into three groups: neuromobilization, tendon gliding, and robotic glove-assisted exercise group.
Who Masked: Outcomes Assessor
Masking Description: All assessments were conducted by a single physiotherapist, who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tendon gliding group (Experimental): The tendon gliding exercises were applied after conventional exercises.
  Interventions: Other: Tendon Gliding Exercise; Other: Conventional Exercises
- Neuromobilization (Experimental): The neuromobilization were applied after conventional exercises.
  Interventions: Other: Neuromobilization Exercise; Other: Conventional Exercises
- Robotic assisted exercises (Experimental): The robotic glove-assisted (RGA) exercise group performed passive movements for 60 minutes using soft robotic gloves (Masmel Health, Turkey), in combination with conventional exercises.
  Interventions: Other: Robotic Assitive Exercise; Other: Conventional Exercises

INTERVENTIONS:
Other: Tendon Gliding Exercise — Tendon gliding exercises were performed for both hands in a sequential manner, with 20 repetitions in 3 sets. The exercises started with fingers and wrist positioned in extension. Subsequent positions included the hook position, full fist position, MCP joint at 90° flexion with finger extension, and MCP and proximal interphalangeal (PIP) joints at 90° flexion positions, with a 5-second hold at each position. During the TG exercises, the hand and fingers are brought to five different positions
  Arms: Tendon gliding group
Other: Neuromobilization Exercise — The neuromobilization exercises included median, radial and ulnar nerve mobilizations. For median nerve mobilization, the patient's wrist was placed in extension, the shoulder in 90° abduction, the forearm in supination, the elbow extended, and the head positioned in lateral flexion toward the same side. For radial nerve mobilization, the wrist was initially placed in flexion and ulnar deviation, the forearm in pronation, with the elbow extended, and the head positioned in lateral flexion toward the same side. For ulnar nerve mobilization, the wrist was positioned in extension and radial deviation, the elbow fully flexed, the forearm in pronation, the shoulder in 90°abduction, and the head in lateral flexion toward the same side. The head was then moved into lateral flexion toward the opposite side while extending the elbow. The neuromobilization protocol was performed in 4 sets of 10 repetitions, with a 5-second hold for each movement.
  Arms: Neuromobilization
Other: Robotic Assitive Exercise — The robotic glove set used in this study weighs 497 grams, powered by a battery weighing 170 grams that provides a 5 V voltage and 1 A current. Made from elastic fabric, the glove wraps around all fingers on both the dorsal and palmar sides. The palm section of the glove is hollow. The device features four Velcro straps: one at the wrist, one across the web space between the thumb and index finger, one between the second and third fingers, and one between the fourth and fifth fingers, securing the inner side of the wrist. The robotic glove facilitates passive joint movements through pneumatic air pressure. The device offers several benefits, including proprioceptive stimulation, visual input, increased functional independence, pain and edema reduction, enhanced lymphatic and blood circulation, improved coordination and hand dexterity, as well as increased grasp and compression strength.
  Arms: Robotic assisted exercises
Other: Conventional Exercises — Wrist extensor exercise, wrist radial deviation exercise, and wrist flexor exercise were perfomed using a 1-kg dumbbell. Holding the 1-kg dumbbell against gravity for 10 seconds, with the shoulder flexed at 90°, elbow extended, and forearm in pronation position. Squeezing exercise with a green soft ball (Thera-Band; diameter: 5 cm); the ball was squeezed for 10 seconds, followed by relaxing. Pushing a blue Pilates ball (Thera-Band; diameter: 20 cm) against the wall with fingers in extension position. Squeezing a black Pilates ring (Thera-Band; diameter: 38 cm) with the fingers, while the MCP joints are in extension and the wrist in a neutral position.

SUMMARY:
The 2018 update of the EULAR recommendations highlighted that exercise reduces pain and improves functionality in patients with hand OA. This study aimed to investigate the effects of neuromobilization, tendon gliding and robotic glove-assisted exercises on pain, grip strength and hand function in patients with hand osteoarthritis (OA).

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic musculoskeletal disorder, and its prevalence increases with age. OA is the most common form of arthritis and is associated with reduced hand functionality and grip strength, increased pain and stiffness, and diminished quality of life. The European League Against Rheumatism (EULAR), the Osteoarthritis Research Society International (OARSI), and the American College of Rheumatology (ACR) have published guidelines for the management of hand OA. The 2018 update of the EULAR recommendations highlighted that exercise reduces pain and improves functionality in patients with hand OA. Previously, strengthening and normal range of motion exercises have been shown to improve grip strength compared to placebo. Moreover, a 2017 Cochrane review reported that interventions involving strengthening, flexibility, stretching, and ROM exercises, either individually or in combination, effectively reduce pain, improve grip strength, alleviate joint stiffness, and enhance functionality in patients with OA.

Among various exercise options, tendon gliding exercises and neuromobilization exercises have been increasingly used in recent years. Neural mobilization aims to restore the balance between neural structures and their surrounding mechanical interfaces, thereby reducing internal neural pressure and facilitating optimal physiological function. When used in combination with conventional treatments, tendon gliding exercises were found to be more effective than nerve gliding exercises in patients with carpal tunnel syndrome.

With technological advancements, the use of robotic assistive devices has become increasingly common in rehabilitation. Robotic devices are primarily used to improve upper limb functionality in neurological conditions, particularly in stroke survivors. These devices assist patients in implementing exercise programs. The use of robotic devices in patients with neurological disorders has been demonstrated to produce positive effects on the central nervous system and sensorimotor deficits. In patients with knee OA, wearable robotic assistive devices have been shown to significantly improve stair-climbing ability and reduce knee pain.

Few studies investigating the efficacy of robotic rehabilitation in hand OA are available in the literature. Research comparing the effects of robotic assistive devices with other treatment methods is still in its early stages. It has been noted by the OARSI that, due to the methodological limitations across studies, and the clinical heterogeneity between studies, it is difficult to provide any reliable practical recommendations for the choice of appropriate therapy in patients with hand OA. Considering the existing gaps in the literature and the recommended research priorities, this study aimed to investigate the effects of neuromobilization, tendon gliding exercises, and the use of a wearable robotic assistive device on pain, grip strength, and hand function in patients with hand OA.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed with primary hand OA by an orthopedics and traumatology specialist based on the ACR diagnostic criteria.
* Aged 45 to 87 years

Exclusion Criteria:

* Individuals were excluded from the study if they had a history of major psychiatric disorders, malignancies, systemic or rheumatologic diseases, severe hand trauma or surgery to the hand region within the past six months, prior intra-articular steroid or hyaluronic acid injections into the hand joints, collagen tissue disorders, peripheral vascular diseases, or a history of neuropathy.

Ages: 45 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Australian-Canadian Hand Osteoarthritis Index | 8 weeks
  The Australian-Canadian Hand Osteoarthritis Index (AUSCAN) is a self-report tool commonly used for the assessment of hand functionality in hand OA. The AUSCAN includes a total of 15 items measuring pain (5 items; 0 to 20 points), stiffness (1 item; 0 to 4 points), and function (9 items; 0 to 36 points) during the preceding 48 hours. Total possible scores range from 0 to 60 points
Jebsen-Taylor Hand Function Test | 8 weeks
  The Jebsen-Taylor Hand Function Test (JTHFT) is used to assess fine and gross motor hand function when performing activities of daily living (ADLs) and to measure the speed at which they perform the test tasks. The JTHFT is a valid and reliable tool and consists of 7 tasks, including writing, turning over cards, picking up objects, stacking checkers, simulated feeding, and moving light and heavy objects. Participants were asked to perform each task separately for each hand, and the time taken for each task was recorded using a stopwatch
Quick Disabilities of the Arm, Shoulder, and Hand (Quick-DASH) questionnaire | 8 weeks
  The Quick-DASH short form consists of a total of 11 questions that ask about an individual's neurological symptoms, pain, sleep disturbances and their ability to work and perform certain activities in the previous week. Each item is assigned a score between 1 and 5: 1 (no difficulty), 2 (mild difficulty), 3 (moderate difficulty), 4 (severe difficulty), 5 (unable). Total possible scores range from 0 (no disability) to 100 (most severe disability). The total score is scaled between 0 (no disability) and 100 (maximum symptoms and disability)
Pain Intensity | 8 weeks
  The Visual Analog Scale (VAS) is a simple, self-administered tool. It consists of a 10-cm line, with the left end representing no pain and the right end representing worst possible pain. Individuals rate their pain intensity by marking a point on VAS, which is scored from 0 to 10.The point marked by the patient on the 10-cm line was measured using a ruler, and the corresponding distance in centimeters was recorded.

SECONDARY OUTCOMES:
Static grip strength | 8 weeks
  A hydraulic hand dynamometer (Jamar, China) was used to measure the static grip strength of the participants. The hydraulic hand dynamometer is a widely used, reliable device for assessing grip strength. Measurements were obtained while the participants were seated upright on a chair, with the MCP joints in a flexion position, elbow flexed at 90°, forearms parallel to the ground, shoulders in adduction, and feet in full contact with the floor. Each measurement was repeated three times, and the highest value in kilograms was noted.
Perceived pain | 8 weeks
  The perceived pain was assessed using the Short-Form McGill Pain Questionnaire (SF-MPQ).The SF-MPQ was designed as a less time-consuming tool than the original MPQ that allows patients to describe their pain intensity in a relatively short period. The tool consists of two subscales with a total of 15 pain descriptors, including 11 sensory descriptors and 4 affective descriptors. Each word is rated on an intensity scale from 0 (none) to 3 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Usgu, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Department of Physiotherapy and Rehabilitation, Gaziantep, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kloppenburg M, Kroon FP, Blanco FJ, Doherty M, Dziedzic KS, Greibrokk E, Haugen IK, Herrero-Beaumont G, Jonsson H, Kjeken I, Maheu E, Ramonda R, Ritt MJ, Smeets W, Smolen JS, Stamm TA, Szekanecz Z, Wittoek R, Carmona L. 2018 update of the EULAR recommendations for the management of hand osteoarthritis. Ann Rheum Dis. 2019 Jan;78(1):16-24. doi: 10.1136/annrheumdis-2018-213826. Epub 2018 Aug 28. PMID 30154087
- [Background] Stoffer-Marx MA, Klinger M, Luschin S, Meriaux-Kratochvila S, Zettel-Tomenendal M, Nell-Duxneuner V, Zwerina J, Kjeken I, Hackl M, Ohlinger S, Woolf A, Redlich K, Smolen JS, Stamm TA. Functional consultation and exercises improve grip strength in osteoarthritis of the hand - a randomised controlled trial. Arthritis Res Ther. 2018 Nov 9;20(1):253. doi: 10.1186/s13075-018-1747-0. PMID 30413191
- [Background] Horng YS, Hsieh SF, Tu YK, Lin MC, Horng YS, Wang JD. The comparative effectiveness of tendon and nerve gliding exercises in patients with carpal tunnel syndrome: a randomized trial. Am J Phys Med Rehabil. 2011 Jun;90(6):435-42. doi: 10.1097/PHM.0b013e318214eaaf. PMID 21430512
- [Background] Mehrholz J, Pohl M, Platz T, Kugler J, Elsner B. Electromechanical and robot-assisted arm training for improving activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2018 Sep 3;9(9):CD006876. doi: 10.1002/14651858.CD006876.pub5. PMID 30175845
- [Background] Pedersini P, Valdes K, Cantero-Tellez R, Cleland JA, Bishop MD, Villafane JH. Effects of Neurodynamic Mobilizations on Pain Hypersensitivity in Patients With Hand Osteoarthritis Compared to Robotic Assisted Mobilization: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2021 Feb;73(2):232-239. doi: 10.1002/acr.24103. Epub 2021 Jan 3. PMID 31675184
- [Background] Villafane JH, Valdes K, Imperio G, Borboni A, Cantero-Tellez R, Galeri S, Negrini S. Neural manual vs. robotic assisted mobilization to improve motion and reduce pain hypersensitivity in hand osteoarthritis: study protocol for a randomized controlled trial. J Phys Ther Sci. 2017 May;29(5):801-806. doi: 10.1589/jpts.29.801. Epub 2017 May 16. PMID 28603349